CLINICAL TRIAL: NCT03259165
Title: Nitroglycerin vs. Furosemide Using Lung Ultrasound Pilot Trial (N-FURIOUS)
Brief Title: Nitroglycerin vs. Furosemide Using Lung Ultrasound Pilot Trial
Acronym: N-FURIOUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19 pandemic. Initially had planned to resume study, but ultimately decided to close.
Sponsor: Indiana University (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, PETER S PANG, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17IRG33411129
Record Dates: First submitted 2017-08-19; First posted 2017-08-23 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure; Heart Failure Acute; Acute Cardiac Failure; Acute Cardiac Pulmonary Edema
Keywords: Heart Failure; Acute Heart Failure; Pulmonary Edema; Lung Ultrasound; Extra vascular lung water; B-lines; Diuretics; Nitrates
MeSH Terms: conditions — Heart Failure; Pulmonary Edema | interventions — Nitrates; Sodium Potassium Chloride Symporter Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrate Intense Strategy (Experimental): Patients randomized to the Nitrate intense strategy will be treated according to protocol with nitrates in combination with IV loop diuretics. This protocol only involves therapies used in everyday AHF clinical practice.
  Interventions: Drug: Nitrates
- Diuretic Intense Strategy (Experimental): Patients randomized to the Diuretic intense strategy will be treated according to protocol with IV loop diuretics in combination with nitrates. This protocol only involves therapies used in everyday AHF clinical practice.
  Interventions: Drug: Loop Diuretics

INTERVENTIONS:
Drug: Nitrates — For patients randomized to the Nitrate intense arm, the treatment protocol will be initiated and continued until there is a decrease in B-lines to ≤ 15 or 6 hours of care has been delivered, whichever comes first.
  Treatment protocol:
  1. IV furosemide (unless already given) (All patients receive at minimum 20 mg IV furosemide or equivalent)
  2. SL nitroglycerin (400 ucg) will be given every 5 minutes, a total of three times. (May be repeated) (Held if SBP decreases to < 120 mmHg)
  3. Reassessment every 2 hours. If LUS B-lines >15, repeat step 2. If < 15, stop algorithm.
  Other Names: SL or IV Nitrates
  Arms: Nitrate Intense Strategy
Drug: Loop Diuretics — For patients randomized to the Diuretic intense arm, the treatment protocol will be initiated and continued until there is a decrease in B-lines to ≤ 15 or 6 hours of care has been delivered, whichever comes first.
  Treatment protocol:
  1. Patients receive 1 inch topical nitropaste
  2. IV Loop diuretic dose = patients total oral dose (max dose of 200 mg IV)
  3. Reassessment every 2 hours. If LUS B-lines >15, repeat step 2. If < 15, stop algorithm.
  Other Names: IV Loop Diuretics
  Arms: Diuretic Intense Strategy

SUMMARY:
Nearly 80% of acute heart failure (AHF) patients admitted to the hospital are initially treated in the emergency department (ED). Once admitted, within 30 days post-discharge, 27% of patients are re-hospitalized or die. Attempts to improve outcomes with novel therapies have all failed. The evidence for existing AHF therapies are poor: No currently used AHF treatment is known to improve outcomes. ED treatment is largely the same today as 40 years ago. Congestion, such as difficulty breathing, weight gain, and leg swelling, is the primary reason why patients present to the hospital for AHF. Treating congestion is the cornerstone of AHF management. Yet half of all AHF patients leave the hospital inadequately decongested.

Although it is the investigators' belief patients are often inadequately decongested in the ED, it is common teaching within emergency medicine to focus on vasodilators and avoid or minimize diuretics, especially in those patients with elevated blood pressure. This practice is largely driven by retrospective analyses or small studies suggesting vasodilators are efficacious and IV loop diuretics may be associated with harm. The evidence base to guide early ED management is poor, and the AHA/ACC guidelines provide little to no guidance for ED treatment. This reflects the lack of high quality data, a critical unmet need that the investigators will address in this study.

Using clearance of LUS B-lines as the study endpoint, the investigators will study whether a diuretic intense vs. nitrate intense strategy achieves better decongestion. Although nearly two decades old, a small study of 100 patients suggested a nitrate intense strategy led to better outcomes in AHF patients with pulmonary edema when compared with a diuretic intense strategy. The investigators aim to perform a small pilot study, in hypertensive patients (SBP > 140mmHg) to test such a strategy to inform a larger, more definitive multicenter randomized trial.

DETAILED DESCRIPTION:
The primary goal of the N-FURIOUS pilot trial is to determine whether a nitrate intense strategy safely reduces congestion, defined by LUS B-lines, better than a diuretic intense strategy.

This pilot trial is designed to provide the necessary and sufficient information for a larger, definitive trial.

PUBLIC HEALTH IMPACT:

Over one million hospitalizations for AHF occur every year in the US. Within 30 days after hospitalization, over 25% of AHF patients will be dead or re-hospitalized. By one year after hospitalization, up to 67% of patients will be re-hospitalized and 36% will be dead. Worldwide, the costs of AHF exceed 100 billion annually. For patients aged 65 years and older, AHF is the most common and most expensive reason for hospitalization. Despite major reductions in morbidity and mortality for chronic HF, considerably less progress has been seen in AHF.

The emergency department (ED) initiates diagnosis and management for the vast majority of AHF patients. Nearly 80% of all admissions originate from the ED. Delays in diagnosis, misdiagnosis, and delayed or improper treatment are costly, associated with greater morbidity and mortality. Despite this crucial starting role, ED AHF pharmacological management today is largely the same as 40 years ago. In fact, guidelines state: "the treatment of AHF remains largely opinion-based with little good evidence to guide therapy." Consensus statements from the American Heart Association as well as a working group from the NHLBI on ED AHF management further corroborate this lack of evidence: "the evidence base on which this foundation of acute care is built is astonishly thin." There remains a critical unmet need for evidence based ED AHF management.

Limitations of Current AHF Therapy:

There are currently no Class I, Level of Evidence A therapeutic guideline recommendations for AHF, highlighting the unmet need. In fact, therapeutic recommendations from the ACCF/AHA begin with hospital based management, highlighting the absence of ED based evidence. The last ED based guidelines were published in 2007 and have yet to be updated. The investigators argue this lack of evidence leads to tremendous variation in ED care. Combined, this contributes to worse outcomes.

Targeting Congestion in AHF:

Freedom from congestion is associated with improved outcomes; yet many patients leave the hospital inadequately decongested. In fact, many patients leave the hospital without a pre-discharge assessment of congestion. The investigators would argue, many ED AHF patients are poorly assessed prior to hospitalization. The absence of robust, reliable methods to assess congestion is a primary reason why it is not assessed. A recent consensus statement published in 2010 highlights this fact: "…no method to assess congestion prior to discharge has been validated." While physical exam is currently the cornerstone of congestion assessment, it lacks sensitivity and inter-rater reliability. The ED is the beginning of AHF management for >75% of admitted patients; delays in diagnosis, misdiagnosis, and resultant delays in management are associated with greater morbidity and mortality.

Initial Therapy:

IV loop diuretics are the mainstay of AHF management. Yet emergency physicians are often reluctant to use IV loop diuretics, largely influenced by small studies and retrospective studies suggesting an association with harm. Nitrates are either recommended above diuretics or even to replace diuretics in popular blogs, podcasts, or online forums. Arguably, neither IV loop diuretics nor nitrates have definitive outcome data regarding efficacy or harm. This is evident in guidelines, where IV loop diuretics receive a class I, B indication, and nitrates a IIb, A recommendation. The evidence that does exist supports their use. Whether one should be used before another, both, how to combine them, and in whom, is not well defined.

Lung Ultrasound as an Endpoint:

For years, the lungs have been considered 'off-limits' to ultrasound: with aerated lungs, the ultrasound beam is reflected and scattered due to acoustic mismatch. However, in the setting of pulmonary congestion, extra vascular lung water (EVLW) can be directly visualized and quantitated. Lung ultrasound measurement of B-lines are an objective, semi-quantitative measure of extra vascular lung water (EVLW). B-lines are well-defined, vertical echogenic lines, originating from water-thickened interlobular septa. They are a marker of congestion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Presents with shortness of breath at rest or with minimal exertion
* Clinical diagnosis of AHF and presence of > 15 total bilateral B-lines distributed in at least 4 zones on initial LUS
* Hx of chronic HF and ANY ONE OF THE FOLLOWING:
* [Chest radiograph consistent with AHF
* Jugular venous distension
* Pulmonary rales on auscultation
* Lower extremity edema
* BNP > 500pg/mL]

Exclusion Criteria:

* Chronic renal dysfunction, including ESRD or eGFR < 20 ml//min/1.73m2.
* Shock of any kind. Any requirement for vasopressors or inotropes.
* SBP < 120
* Need for immediate intubation
* Acute Coronary Syndrome OR new ST-segment elevation/depression on EKG. (troponin release outside of ACS is allowed)
* Fever >101.5ºF
* End stage HF: transplant list, ventricular assist device
* Anemia requiring transfusion
* Known interstitial lung disease
* Suspected acute lung injury or acute respiratory distress syndrome (ARDS)
* Pregnant or recently pregnant within the last 6 months
* Severe valvular disease
* Anuria
* Allergy or hypersensitivity to nitroglycerin, furosemide or sulfa
* Concern for cardiac tamponade or restrictive cardiomyopathy
* Elevated intracranial pressure
* Recent use of PDE5 inhibitors

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Pang, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Eskenazi Health, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitrate Intense Strategy: Patients randomized to the Nitrate intense strategy will be treated according to protocol with nitrates in combination with IV loop diuretics. This protocol only involves therapies used in everyday AHF clinical practice.
  Nitrates: For patients randomized to the Nitrate intense arm, the treatment protocol will be initiated and continued until there is a decrease in B-lines to ≤ 15 or 6 hours of care has been delivered, whichever comes first.
  Treatment protocol:
  1. IV furosemide (unless already given) (All patients receive at minimum 20 mg IV furosemide or equivalent)
  2. SL nitroglycerin (400 ucg) will be given every 5 minutes, a total of three times. (May be repeated) (Held if SBP decreases to < 120 mmHg)
  3. Reassessment every 2 hours. If LUS B-lines >15, repeat step 2. If < 15, stop algorithm.
- Diuretic Intense Strategy: Patients randomized to the Diuretic intense strategy will be treated according to protocol with IV loop diuretics in combination with nitrates. This protocol only involves therapies used in everyday AHF clinical practice.
  Loop Diuretics: For patients randomized to the Diuretic intense arm, the treatment protocol will be initiated and continued until there is a decrease in B-lines to ≤ 15 or 6 hours of care has been delivered, whichever comes first.
  Treatment protocol:
  1. Patients receive 1 inch topical nitropaste
  2. IV Loop diuretic dose = patients total oral dose (max dose of 200 mg IV)
  3. Reassessment every 2 hours. If LUS B-lines >15, repeat step 2. If < 15, stop algorithm.
Period: Overall Study
Arm/Group | Nitrate Intense Strategy | Diuretic Intense Strategy
Started | 27 | 25
Completed | 26 (Study halted prematurely due to COVID-19. Patient lost to follow up) | 24 (Study halted prematurely due to COVID-19 pandemic. Patient lost to follow up)
Not Completed | 1 | 1
Not completed — COVID 19 pandemic | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrate Intense Strategy | Diuretic Intense Strategy | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 23 | 19 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 15 | 26
  White | 15 | 10 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: The Total Number of B-lines at the Conclusion of ED AHF Management
Description: The total number of B-lines at the conclusion of ED AHF management or maximum of 6 hours after enrollment, whichever comes first.
Time Frame: During the ED phase of management, no more than 6 hours
Population: The trial was halted prematurely because of the COVID-19 pandemic. There is insufficient funding for data to be analyzed properly, at the time of this submission. Of the original 52 patients, only 9 in the Nitrate Arm and 7 in the Diuretic Intense arm had reported data of a LUS performed at the completion of ED treatment (t6)
Measure: Mean (Standard Deviation); unit: Number of B-lines
Arm/Group | Nitrate Intense Strategy | Diuretic Intense Strategy
Number analyzed (Participants) | 9 | 7
Number of B-lines | 29 (22.5) | 32 (19.4)

2. Secondary Outcome: Dyspnea Assessment
Description: A patient reported measurement of dyspnea using 7-point Likert scales in a standardized position, ranging from Markedly worse, Moderately Worse, Minimally Worse, No Change to Minimally Improved, Moderately Improved, Markedly Improved
Time Frame: During the ED phase of management, no more than 6 hours
Population: • The trial was halted prematurely due to the COVID-19 pandemic. There is insufficient funding for data to be analyzed properly at the time of this submission. Only 15 patients had data available to report
Measure: Number; unit: participants
Arm/Group | Nitrate Intense Strategy | Diuretic Intense Strategy
Number analyzed (Participants) | 10 | 5
participants
  Markedly Improved | 3 | 1
  Moderately Improved | 1 | 3
  Minimally Improved | 4 | 0
  No Change | 1 | 1
  Minimally Worse | 1 | 0

3. Secondary Outcome: B-lines <= 15 at the Conclusion of ED AHF Management
Description: B-lines <= 15 at the conclusion of ED AHF management or maximum of 6 hours after enrollment, whichever comes first
Time Frame: During the ED phase of management, no more than 6 hours
Population: • The trial was halted prematurely due to the COVID-19 pandemic. There is insufficient funding for data to be analyzed properly at the time of this submission. Only 16 patients had reported data for this endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | Nitrate Intense Strategy | Diuretic Intense Strategy
Number analyzed (Participants) | 9 | 7
Participants | 2 | 0

4. Other Pre Specified Outcome: Total DAOOH
Description: Total days alive and out of hospital through 30 days post-discharge
Time Frame: Up through 30 days post discharge
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Association of B-lines at Discharge and 30-day Outcome
Time Frame: Up through 30 days post discharge
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Time to Reach B-lines <15
Time Frame: Throughout hospitalization, on average 5-7 days
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Association of Baseline, Discharge, and Change of B-lines With 30-day Outcomes
Time Frame: Up through 30 days post discharge
Reporting Status: Not Posted

8. Other Pre Specified Outcome: All Cause Readmissions, All Cause ED Re-visits
Time Frame: 30 days post discharge
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Physical Exam Findings and Body Weight From Presentation to Pre-discharge
Description: Physical exam includes peripheral edema, jugular venous distention, pulmonary and cardiac auscultation
Time Frame: From admission to pre-discharge from the hospital, on average 5 to 7 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The study period during which AEs must be reported begins after informed consent is obtained and initiation of study treatment and for 5 days after ending study treatment. Patients will be followed for 30 days for ED visits, re-hospitalization, and mortality. Subject's hospital discharge summaries will be examined at hospital discharge and all non-exempt AEs will be investigated by examining necessary medical records.
Arm/Group | Nitrate Intense Strategy | Diuretic Intense Strategy
All-Cause Mortality (participants affected / at risk) | 1/27 | 2/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/25
Other Adverse Events (participants affected / at risk) | 3/27 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrate Intense Strategy (N=27) | Diuretic Intense Strategy (N=25)
Death (Cardiac disorders) | 0 (0) | 1 (1) — Unknown True Organ System. Death was recorded within 5 days of AE reporting period, however, not cause of death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrate Intense Strategy (N=27) | Diuretic Intense Strategy (N=25)
CTCAE (Renal and urinary disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, enrollment was halted. The nature of the study was to enroll patients with AHF signs and symptoms. The principle symptom is shortness of breath, a common symptom during the peak of COVID-19. Further, employees were not allowed into the ED setting to enroll patients, when much less was known about COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT03259165/Prot_SAP_000.pdf